CLINICAL TRIAL: NCT03667885
Title: Non-Invasive Diagnostics of Small Renal Masses
Acronym: NISar
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Anders Ullmann Kiis Frey, Principal investigator, Odense University Hospital
Other Study IDs: OP_125
Record Dates: First submitted 2018-08-01; First posted 2018-09-12 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Renal Cell Carcinoma; Renal Tumor
Keywords: next generation sequencing; multi planar magnetic resonance; liquid biopsies; non-invasive diagnostics; biomarkers
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — Blood, urine, and tumor samples will be collected and analysed for an array of mRNAs and DNA biomarkers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Small renal Masses: patients with a renal mass of 4 cm or less. Typically incidentally found. Blood and urine samples will be collected from each patient at baseline before a biopsy of the tumor is collected and 14 days later. In addition, all patients will be offered a Multi planar MRI before the biopsy. Patients elected for curative treatment for malignant tumors will have another set of blood and urine samples collected at 1 month and 6 months after the intervention.
  Interventions: Diagnostic Test: Blood sample; Diagnostic Test: urine sample; Diagnostic Test: Multi planar MRI

INTERVENTIONS:
Diagnostic Test: Blood sample — basic blood sample
Diagnostic Test: urine sample — basic urine sample
Diagnostic Test: Multi planar MRI — T1 (with reduced affinity for fatty tissue) +/- contrast, diffusion weighted sequences and wash in/wash out

SUMMARY:
NiSAR is a Ph.D. study and consists of three substudies. Renal cancer is one of the most deadly urologic malignancies and accounts for 900 new cases and 300 deaths per year. An increase in the use of imaging diagnostics has yielded a rise in the incidental detection of small renal masses (SRM), meaning tumors <4cm (T1a). Kidney biopsies are the gold standard for diagnosing SRM but has an inherent risk of infections, retroperitoneal bleeding and in rare cases loss of kidney function. This is problematic since up to 30% of SRM are benign.

This Ph.D. consists of three studies that all aim to develop new minimally invasive modalities for diagnosing SRM. Patients eligible for these studies are diagnosed with SRM at one of the departments of Urology in the southern region of Denmark. Studies 1 and 2 aims to find circulating biomarkers, in the form of DNA and messenger ribonucleic acid (mRNA) contained in micro vesicles secreted into blood by renal cell cancers and find changes in biomarkers levels after surgery. Study 3 aim to determine the potential of multiplanar MRI (mpMRI) to discriminate between benign and malign SRM. Potentially this can lead to a fundamental change of the way urologists diagnose and monitor SRM and renal cell cancer in general.

The investigators will also build a research biobank for future research.

DETAILED DESCRIPTION:
Study 1:

Trial objective:

Identification of biomarkers in blood and urine and to set the basis for a minimally invasive diagnostic program for SRM.

Method:

Sample collection:

All blood samples will be collected in ethylendiamin-tetraacetate (EDTA) containing tubes. two samples are then centrifugated at 2000 G for 10 minutes to isolate plasma, which then are stored at -80oC. The remaining 2 samples are stored at -80oC as is. Total nucleic acid (TNA) will be extracted from concentrated urine and plasma samples as previously described using a NucliSENS easy MAG instrument. Extracted TNA will then be used for targeted immune- and oncologic profiling (mutations and expression) using next generation sequencing (NGS)-based RNA and DNA sequencing.

The additional core sample from kidney tumor will be stored without preservatives for NGS-based DNA and RNA-seq analysis.

Study 2:

Trial objective:

Identification of changes in circulating biomarkers after curative treatment in patients with biopsy verified renal cancer.

Methods:

Patient recruitment:

Patients will be enrolled in study 2 in the same manner as study 1.

Sample collection:

In addition to the first four samples four additional blood samples (20 ml) will be taken 1 month and 6 months after curative treatment from each patient. All samples will be coded and given an ID according to patient´s CPR number using the RedCap informatic coding system.

Sample storage, preparation and analysis:

Blood and urine samples will be handled in the same manner as in study 1. Statistical Analysis for study 1 and 2:

Exploratory analysis of the data will be performed on molecular expression levels of specific sequences identified, an unsupervised hierarchical clustering will be fit and heat maps will be produced. Properties of clustered elements will be further matched with histopathological results to search for histological aggregation patterns.

Expression levels of the sequences identified, in blood and urine will be compared by means of Whitney U test and Kruskal-Wallis test. Changes in levels of expression from pre-operative to post-operative will be evaluated with Friedman´s ANOVA and subsequent post-hoc pairwise comparison with Wilcoxon's signed rank test with Bonferroni correction.

Receiver operating characteristic curve analysis will be further performed on pre-operative samples, to test for validity of the assays for each marker to discriminate between benignant histology and malignancy, with a cut-off for area under curve (AUC) of 0.75.

Sample size The minimal sample size required for achieving a statistical power of 80% with a significance level of 0.05 and an expected dropout rate of 15% will be 155 patients.

Calculations for sample size have been computed with the GPower software (Düsseldorf, DE).

Study 3:

Trial objective:

To investigate the diagnostic value of mpMRI in determining malignancy in SRM.

Method:

Patient recruitment:

After providing a written consent a mpMRI will be scheduled at the same day but prior to the primary biopsy. All mpMRIs will be performed locally and the pictures transferred to Odense University Hospital where a specialist radiologist, will examine the scans in a blinded fashion, meaning that he will be ignorant to the pathologist´s diagnosis. The result will be stored in a coded RedCAP database.

MpMRIs are performed according to a standard protocol and include the following sequences: T1 (with reduced affinity for fatty tissue) +/- contrast, diffusion weighted sequences and wash in/wash out.

ELIGIBILITY:
Inclusion Criteria:

* All patients with SRM < 4cm (T1a) at the Departments of Urology in the region of Southern Denmark.
* Written consent
* Able to speak and understand Danish

Exclusion Criteria:

* Patients below 18 years of age,
* Patients with mental impairment
* Withdrawal of consent
* Other malignancies.

Specific for study 2:

* Patients unsuitable for curative treatment.

Specific for study 3:

* Pregnancy
* Kidney failure
* Kidney-grafts
* History of allergic-reactions to contrast agents
* Patients with non-MRI-compatible components
* Patients unable to cooperate for an MRI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who presents with a small renal mass <4cm.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Expression of mRNA and DNA markers | Baseline
  Expression levels of the sequences identified, in blood and urine will be compared by means of Whitney U test and Kruskal-Wallis test.
Change in mRNA and DNA markers | 1 month, and 6 months
  Changes in levels of expression from pre-operative to post-operative will be evaluated with Friedman´s ANOVA and subsequent post-hoc pairwise comparison with Wilcoxon's signed rank test with Bonferroni correction
Analysis of MpMRIs | Baseline
  A specialist radiologist will examine the scans in a blinded fashion, meaning that he will be ignorant to the pathologist´s diagnosis.

SECONDARY OUTCOMES:
Expression of mRNA and DNA markers | Fourteen days after first samples
  Expression levels of the sequences identified, in blood and urine will be compared by means of Whitney U test and Kruskal-Wallis test.

CONTACTS AND LOCATIONS:
Overall Officials: Anders U Frey, Ph.D student, Principal Investigator — Odense UH
Locations (1):
- Odense Universitets Hospital, Odense, Fyn, Denmark

IPD SHARING:
Plan to Share IPD: No